CLINICAL TRIAL: NCT04946097
Title: Effect of Gross Myofascial Release on Pain and Function in Cervical Radiculopathy Patients: A Randomized Controlled Study
Brief Title: Gross Myofascial Release in Cervical Radiculopathy Pat
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Lama Saad El-Din Mahmoud, Lecturer of physical therapy, Department of Neuromuscular disorders and its surgery, faculty of physical therapy, october 6 univerisity, October 6 University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T. REC/012/003223
Record Dates: First submitted 2021-06-22; First posted 2021-06-30 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Cervical Radiculopathy
MeSH Terms: conditions — Radiculopathy | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: the control group which received the conventional selected exercise program and the study group received the same exercise training program in addition to gross Myofascial Release
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): received the conventional selected exercise program in addition to gross Myofascial Release
  Interventions: Other: gross Myofascial Release; Other: conventional selected exercise program; Device: Transcutaneous electrical nerve stimulation (TENS)
- control group (Experimental): the control group which received the conventional selected exercise program
  Interventions: Other: conventional selected exercise program; Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Other: gross Myofascial Release — Gross Myofascial Release : is amanual technique in form of Stretch of the Posterior Cervical Musculature and Gross stretch of gross Myofascial Release upper quarter: Arm Pull for duration of 10-15 min per session each stretch position was healed for 90sec
  Arms: study group
Other: conventional selected exercise program — stretching exercises for cervical muscles and pectoralis major and source of heat in form of hot packs for 15 minutes
Device: Transcutaneous electrical nerve stimulation (TENS) — Transcutaneous electrical nerve stimulation (TENS) is a method of pain relief involving the use of electrical current, the electrode placement on the course of pain for 15 minutes
  Other Names: TENS

SUMMARY:
To investigate the Effect of gross Myofascial Release on pain and function in cervical radiculopathy patients. BACKGROUND: cervical radiculopathy is considered serious problems causing neck pain & radiating pain which affect physical inactivity and function of a patient, thus gross Myofascial Release is a form of manual therapy technique that has a profound effect upon the musculoskeletal system.

HYPOTHESES:

This study hypothesized that:

gross Myofascial Release on pain and function in cervical radiculopathy patients RESEARCH QUESTION: Is there an effect of gross Myofascial Release on pain and function in cervical radiculopathy patients?

DETAILED DESCRIPTION:
Forty patients with cervical radiculopathy will participate in this study. The patients will randomly be divided into two equal groups; the control group which received the conventional selected exercise program and the study group received the same exercise training program in addition to gross Myofascial Release, three times per week for four weeks. The evaluation methods are visual analogue scale (VAS), Electro-goniometer, Quick DASH scale, and Neck disability index

ELIGIBILITY:
Inclusion Criteria:

* 40 cervical radiculopathy patients,
* Age will range as (30:45) years old
* Cervical radiculopathy due to cervical spondylosis
* body mass index (25:29)

Exclusion Criteria:

* difficulty to communicate or to understand program instructions
* any other neurological deficits or orthopaedic abnormalities,
* secondary musculoskeletal complication
* Cervical disc prolapses
* Any other cervical problem
* Spinal stenosis
* Previous spinal surgery

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Electro-goniometer | 4 weeks
  Measurement of cervical range of motion in four direction flexion, extension side bending and rotation
Quick Disabilities of the Arm, Shoulder and Handscale | 4 weeks
  The Quick Disabilities of the Arm, Shoulder and Hand (DASH) scale only contains 11 items, It is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. The Quick Disabilities of the Arm, Shoulder and Hand tool uses a 5-point Likert scale from which the patient can select an appropriate number corresponding to his/her severity/function level, as the higher scores indicate a greater level of disability and severity, whereas, lower scores indicate a lower level of disability, and The score ranges from 0 (no disability) to 100 (most severe disability)
Neck Disability Index | 4 weeks
  The Neck Disability Index is designed to measure neck-specific disability. The questionnaire has 10 items concerning pain and activities of daily living including personal care, lifting, reading, headaches, concentration, work status, driving, sleeping and recreation. The measure is designed to be given to the patient to complete, and can provide useful information for management and prognosis of those with neck pain.The test maximum score of 50, or as a percentage. as 0 points or 0% means : no activity limitations , and 50 points or 100% means complete activity limitation.
  A higher score indicates more patient-rated disability.

SECONDARY OUTCOMES:
visual analogue scale | four weeks
  for the assessment of the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain. The most simple visual analogue scale is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the degree of pain to be measured, as the higher scores (100mm) indicate a greater intensity of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Hosam M Metwally, PHD, Principal Investigator — lecturer , department of Neuromuscular Disorders and its surgery, faculty of physical therapy O6U physical therapy; Lama Saad ED Mahmoud, PHD, Study Chair — October 6 University; Sobhy M Aly, PHD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - October 6 university, Giza, Giza Governorate
  - October 6 university, Al Jīzah, Select State